CLINICAL TRIAL: NCT01181336
Title: A Single Centre, Randomised, Double Blind, Phase 1 Study of the Safety, Tolerability, and Immunogenicity of an Influenza Vaccine Candidate (FLU-v)
Brief Title: Phase 1b Influenza Vaccine Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepTcell Limited (Industry)
Responsible Party: Dr. Stuart Robinson, PepTcell Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU-v-001
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Influenza
Keywords: Safety; Tolerability; Immunogenicity; Influenza; Virus; Vaccine
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 2 (Experimental): FLU-v Low Dose with adjuvant. FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences). Administration: A single subcutaneous injection.
  10 subjects.
  Interventions: Biological: Influenza vaccine (FLU-v)
- Group 3 (Experimental): FLU-v High Dose with water for injection. FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences). Administration: A single subcutaneous injection.
  10 subjects.
  Interventions: Biological: Influenza vaccine (FLU-v)
- Group 4 (Experimental): High Dose FLU-v with adjuvant FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences). Administration: A single subcutaneous injection. 10 subjects
  Interventions: Biological: Influenza vaccine (FLU-v)
- Group 1 (Experimental): FLU-v Low Dose with water for injection FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences). Administration: A single subcutaneous injection 10 subjects
  Interventions: Biological: Influenza vaccine (FLU-v)
- Control Group (Placebo Comparator): Placebo with adjuvant (4 subjects) or Placebo without adjuvant (4 subjects)
  Interventions: Biological: FLU-v Control

INTERVENTIONS:
Biological: Influenza vaccine (FLU-v) — Comparison of different dosages of FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences). Administration: A single subcutaneous injection of (Low Dose / High Dose with adjuvant / water for injection)
  Other Names: FLU-v
  Arms: Group 1; Group 2; Group 3; Group 4
Biological: FLU-v Control — Adjuvant only or water for injection only Administration: a single subcutaneous injection
  Arms: Control Group

SUMMARY:
The purpose of this study is to see whether a single vaccination (injection) with the investigational influenza vaccine is safe in healthy subjects. The study is also designed to evaluate four different dose formulations of the vaccine to see which gives the best immune response.

DETAILED DESCRIPTION:
Prophylactic vaccination against influenza is indicated for "at risk" populations including patients suffering from chronic respiratory diseases (including asthma), chronic heart disease, chronic renal failure, diabetes mellitus and immunosuppression due to disease or treatment. Vaccination of the elderly (>65 years) and the residents of nursing homes is also recommended. The current influenza vaccines available contain subunits from two influenza A viruses and an influenza B virus and consist either of inactivated whole virus or subunits of haemagglutinin and neuraminidase.

The investigational influenza vaccine (FLU-v) contains multiple highly conserved T cell epitopes that are present on most influenza viruses, which have been identified as reactive in different human leukocyte antigen (HLA) populations; thus making it unlikely that anybody in the vaccinated population would be unable to mount an immune response to at least one of the epitopes contained in the vaccine.

This study will be the initial exploration of FLU-v in humans, and aims to assess the safety, tolerability, and immunogenicity in healthy subjects.

Subjects will be randomised to receive either Low Dose or High Dose FLU-v with or without adjuvant, or placebo with or without adjuvant. Twenty-four (24) subjects will be randomized to Low Dose and 24 subjects to High Dose. To mitigate risk, a staggered dosing approach will be used. One subject will receive Low Dose FLU-v without adjuvant, and one subject will receive placebo without adjuvant, followed 6 hours later by one subject receiving Low Dose FLU-v with adjuvant, and one subject receiving placebo with adjuvant. All 4 subjects will be observed overnight. At least 72 hours later and in the absence of any clinically-significant safety signals (as determined by a Safety Review Committee) the remaining 20 subjects of the Low Dose group will be dosed. If deemed appropriate by the Safety Review Committee a second sentinel cohort of 4 subjects will be observed overnight prior to completing the remaining subjects of the Low Dose group. Following a satisfactory review of safety data from the combined Low Dose cohorts, subjects in the High Dose group will be vaccinated using the same staggered dosing approach as used in Low Dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a BMI >18.5 and ≤ 28.5 kg/m2.
* Subject must have no clinically significant abnormal findings, as judged by the Investigator, on the physical examination, ECG, medical history or clinical laboratory results during screening.
* Subject must be a non-user of tobacco products, or smoke ≤ 10 cigarettes per day (minimum 6 months prior to first dose).
* Subject must have a negative urine screen for drugs of abuse and a negative alcohol breath test at screening and check-in.
* Subject must refrain from consuming alcohol for 72 hours prior to each dose.
* Subject must be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator.
* Subject must give voluntary written informed consent to participate in this trial.

Exclusion Criteria:

* Subject must not have previous influenza vaccination within the 12 months prior to test drug vaccination.
* Subject must not have had an influenza like illness within the 3 months prior to test drug vaccination.
* Subject must not have a history or presence of significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, haematological or renal disorder.
* Subject must not have an oral temperature >38°C on day of vaccination (otherwise subject maybe be re-assigned to a subsequent cohort).
* Subject must not suffer from an inherited or acquired immunodeficiency.
* Subject must not suffer from a disease or be undergoing treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800µg/day beclometasone or equivalent), radiation treatment, cytotoxic drugs or non-steroidal anti-inflammatory drugs.
* Subject must not have a serologically positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Subject must not have a history of severe allergic reactions and/or anaphylaxis.
* Subject must not have any arm rash or tattoos which could confound the interpretation of any injection site reactions.
* Subject must not have participated in a previous clinical trial within 90 days prior to the first vaccination.
* Subject must not have donated blood or plasma more within 90 days prior to the first vaccination.
* Subject must not have donated bone marrow within 6 months prior to the first dose.
* Subject must not have received administration of immunoglobulins and/or any blood products within 90 days prior to the first vaccination, or any planned administration during the study period.
* Subject must not use any prescription medication within 14 days prior to the first vaccination.
* Subject must not use over-the-counter (OTC) medication 7 days prior to the first vaccination. Exceptions are described below under the heading 9.4.1.
* Subject must not have received any vaccine within the 30 days prior to the first dose, and must agree not to receive any other vaccine (other than any vaccine indicated for standard of care, for example, tetanus vaccine) for the duration of this study i.e 21 days post initial FLU-v vaccination.
* Subject must not have a history of alcohol or drug abuse within 2 years prior to the first dose.
* Subject must not have any condition which, in the judgement of the Investigator, precludes inclusion into the study.
* Subjects must not donate sperm up to 90 days postdose, and those whose partner is of child-bearing potential will be advised to remain sexually inactive or use a dual method of birth control (e.g. condom together with spermicidal agent, IUD or hormonal contraception) for at least 90 days postdose.
* Subject must not be a direct employee of the study site, monitoring CRO or Sponsor.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of FLU-v | Measurements will be taken at screening, then up to 21 days post-vaccination
  The safety and tolerability of two dose levels of FLU-v and the effect of the adjuvant on the safety and tolerability of FLU-v will be assessed by, Clinical signs and symptoms from physical exam and ECG; Adverse events (including local and systemic AEs); Laboratory safety (haematology, serum clinical chemistry, urinalysis); and Vital signs (blood pressure, heart rate, temperature, respiratory rate)

SECONDARY OUTCOMES:
Immunogenicity of FLU-v | Measurements will be taken on Days 1 and 21 post-vaccination
  The immunogenicity of FLU-v with and without adjuvant will be measured by Serum IgG2 (assessed by enzyme-linked immunosorbant assay (ELISA)) and IFN-γ in isolated peripheral blood mononuclear cells (PBMC).

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Robinson, Dr, Study Director — PepTcell Limited
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Pleguezuelos O, Robinson S, Stoloff GA, Caparros-Wanderley W. Synthetic Influenza vaccine (FLU-v) stimulates cell mediated immunity in a double-blind, randomised, placebo-controlled Phase I trial. Vaccine. 2012 Jun 29;30(31):4655-60. doi: 10.1016/j.vaccine.2012.04.089. Epub 2012 May 8. PMID 22575166